CLINICAL TRIAL: NCT02541240
Title: Effects of an Intervention to Enhance Resilience in Physical Therapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Responsible Party: Principal Investigator, Anne Mejia-Downs, Principal Investigator, University of Indianapolis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RARMUoHP063015
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Psychological Stress
Keywords: resilience; optimism; stress; coping; curriculum
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resilience Curriculum (Experimental): The intervention is exposure to an 8-hour Resilience Curriculum. It will provide education for participants about methods to increase protective factors against stress, the use of effective coping strategies, and the importance of accessing social support, with the goal of better managing stress and enhancing resilience. The curriculum will include a didactic component, skills-building training, and homework exercises to encourage the application of the skills.
  Interventions: Other: Resilience Curriculum
- No Resilience Curriculum (No Intervention): The Waitlist Control group will receive no exposure to the Resilience Curriculum. After the final data is collected, this group will be offered the opportunity to attend a condensed 2-hour version of the curriculum.

INTERVENTIONS:
Other: Resilience Curriculum — The Resilience Curriculum consists of 4 modules, with one 2-hour module presented each week.
  Arms: Resilience Curriculum

SUMMARY:
Health professional students experience high levels of psychological stress. Individuals with higher levels of resilience are better equipped to handle stress. The purpose of this study is to evaluate the effects of an 8-hour resilience curriculum on stress levels, resilience, coping, protective factors, and symptomatology on students enrolled in a doctor of physical therapy (DPT) program.

Hypothesis: The curriculum will decrease stress levels, increase resilience, coping flexibility, protective factors (optimism, positive affect, and social support), and reduce symptomatology (negative affect, illness). Research on stress and its consequences experienced by physical therapy students in particular is limited. If the results of this study support this hypothesis, it may establish the benefit of adding a resilience component to the curriculum for students of physical therapy.

DETAILED DESCRIPTION:
The study involves curriculum development and evaluation by randomized controlled trial. Participants will be randomized to the intervention group to receive a Resilience Curriculum or to a wait-list control group to receive a condensed version of the curriculum following the post-intervention assessments.

Pre- and post-intervention assessments will be administered to both groups, with baseline assessments administered in the first two weeks of the semester. The assessments will include measures of stress levels, levels of resilience, coping flexibility, optimism, positive and negative emotions, social support, and symptoms of illness. The intervention, the presentation of a resilience curriculum, will be delivered to the intervention group during the week following the baseline assessments and it will last for four weeks.

The resilience curriculum will provide education for participants about methods to increase protective factors against stress, the use of effective coping strategies, and the importance of accessing social support, with the goal of better managing stress and enhancing resilience. The intervention will include a didactic component, skills-building training, and homework exercises to encourage the application of the skills. The curriculum will be delivered in four 2-hour modules, with one module delivered each week. The follow-up assessments will occur after midterm examinations are concluded. An abbreviated curriculum which will last approximately two hours will be delivered to the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Current enrollment in Doctor of Physical Therapy program at either Indiana University or the University of Indianapolis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in psychological resilience at 8 weeks | Baseline and 8 weeks
  The 25-item Connor-Davidson Resilience Scale measures a variety of constructs of resilience including hardiness, personal competence, social bonds, patience, and spiritual influences.

SECONDARY OUTCOMES:
Change from baseline in perceived psychological stress at 8 weeks | Baseline and 8 weeks
  The 10-item Perceived Stress Scale was created to assess the perception of stress in the previous month,
Change from baseline in coping flexibility at 8 weeks | Baseline and 8 weeks
  The Coping Flexibility Scale is a 10-item tool to measure the ability of an individual to effectively modify coping behavior.
Change from baseline in optimism at 8 weeks | Baseline and 8 weeks
  The Revised Life Orientation Test is a 10-item scale designed to measure optimism in an individual.
Change from baseline in positive and negative emotions at 8 weeks | Baseline and 8 weeks
  The 20-item Modified Differential Emotion Scale, an adaptation of the original Differential Emotion Scale, measures positive and negative emotions that an individual has experienced in the previous 2 weeks.
Change from baseline in social support at 8 weeks | Baseline and 8 weeks
  The Social Provisions Scale is a 24-item assessment of six areas of social relationships (guidance, reliable alliance, attachment, social integration, reassurance of worth, and opportunity for nurturance) used to measure perceived social support.

OTHER OUTCOMES:
Change from baseline in symptoms of Illness at 8 weeks | Baseline and 8 weeks
  The Symptoms of Illness Checklist is a 33-item tool designed to measure the number, frequency, and severity of physical symptoms experienced in the previous two-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Mejia-Downs, PT, MPH, Principal Investigator — University of Indianapolis
Locations (2):
- United States (2):
  - Indiana University Purdue University Indianapolis, Indianapolis, Indiana
  - University of Indianapolis, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared.

REFERENCES:
- [Background] O'Leary VE, Ickovics JR. Resilience and thriving in response to challenge: an opportunity for a paradigm shift in women's health. Womens Health. 1995 Summer;1(2):121-42. PMID 9373376
- [Background] Walsh JM, Feeney C, Hussey J, Donnellan C. Sources of stress and psychological morbidity among undergraduate physiotherapy students. Physiotherapy. 2010 Sep;96(3):206-12. doi: 10.1016/j.physio.2010.01.005. Epub 2010 Apr 8. PMID 20674652
- [Background] Jacob T, Itzchak EB, Raz O. Stress among healthcare students--a cross disciplinary perspective. Physiother Theory Pract. 2013 Jul;29(5):401-12. doi: 10.3109/09593985.2012.734011. Epub 2012 Oct 24. PMID 23094641
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Tugade MM, Fredrickson BL. Resilient individuals use positive emotions to bounce back from negative emotional experiences. J Pers Soc Psychol. 2004 Feb;86(2):320-33. doi: 10.1037/0022-3514.86.2.320. PMID 14769087
- [Background] Steinhardt M, Dolbier C. Evaluation of a resilience intervention to enhance coping strategies and protective factors and decrease symptomatology. J Am Coll Health. 2008 Jan-Feb;56(4):445-53. doi: 10.3200/JACH.56.44.445-454. PMID 18316290
- [Background] McAllister M, McKinnon J. The importance of teaching and learning resilience in the health disciplines: a critical review of the literature. Nurse Educ Today. 2009 May;29(4):371-9. doi: 10.1016/j.nedt.2008.10.011. Epub 2008 Dec 3. PMID 19056153
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174